CLINICAL TRIAL: NCT03769909
Title: Inhibition of Inflammation for Prevention of Posttraumatic Osteoarthritis After Acute Intraarticular Fractures
Brief Title: Prevention of Posttraumatic Osteoarthritis After Acute Intraarticular Fractures
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: University of Freiburg (Other); Odense University Hospital (Other); The Danish Rheumatism Association (Other); Hartmann Fonden (Other); AP Møller Fond (Unknown)
Responsible Party: Sponsor
Other Study IDs: S-20170139
Record Dates: First submitted 2018-11-09; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Ankle Fractures; Intra-Articular Fractures; Osteoarthritis
Keywords: PTOA; Osteoarthritis; Intra-Articular Fractures; Ankle Fractures; Cytokines; Biomarkers; Inflammation; Pro-inflammatory; Cartilage; Fracture; Joint Injury
MeSH Terms: conditions — Ankle Fractures; Intra-Articular Fractures; Osteoarthritis; Inflammation; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (5.0-20.0 ml) Synovial Fluids (1.0-10.0 ml) from both ankle joints
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intra-articular fracture is a very common fracture. The only method to treat these fractures is surgery with plate and screws followed by rehabilitation. Even though the surgeons do their best to restore the anatomy, up to 40 percent of the patients develop osteoarthritis after 10 years. Previous research has shown that immediately after fracture in the joint, the body starts an inflammatory response and activates a series of biomarkers inside the joint space. Some of these biomarkers are believed to break down the cartilage resulting in development of osteoarthritis, despite surgical treatment. Currently it is still unknown, which biomarkers are activated in the joint space, and how we can stop their deleterious action in order to prevent cartilage degradation.

The purpose of this project is to identify the biomarkers in the joint space after an intra-articular ankle fracture and to evaluate how these biomarkers affect the short- and mid-terms clinical outcomes. As secondary outcomes we evaluate how fracture classification and fracture reduction affect clinical outcomes and physical activity after surgery.

DETAILED DESCRIPTION:
Osteoarthritis (OA) affecting one in eight individuals and is the main reason for chronic pain and disability worldwide. The main cause for OA development is joint-affecting trauma and risk factors have primarily been associated to previous biomechanical treatment. Therefore, the principle of current fracture treatment is anatomical reconstruction of the joint surface combined with functional and adequate aftercare. However, despite correct restoration of anatomy and application of sufficient physiotherapy, the risk of posttraumatic OA remains as high as 40%.

Joint trauma initiates an inflammatory cascade leading to synovial catabolism and cartilage degradation, a fact, which to date has been ignored in standard therapy. Unfortunately, due to the lack of blood supply, cartilage regenerates much less efficient compared to bone. Previous studies suggest that the synovial biochemical milieu may be of decisive importance for chondrocyte and cartilage survival or degeneration. The investigators therefore hypothesize, that protecting cartilage and chondrocyte by inhibiting the post-injury inflammatory cascade, might contribute to durable successful results in fracture therapy. The purpose of this project is to identify the biomarkers in the joint space after an intra-articular ankle fracture and to evaluate how these biomarkers affect the short- and mid-terms clinical outcomes. As secondary outcomes we evaluate how fracture classification and reduction affect clinical outcomes and physical activity after surgery. In specific, we intend to answer the following research questions:

Study 1: Are there differentially regulated biomarkers in joint space in patients with and without an intra-articular ankle fracture?

Study 2: Do the identified biomarkers found in intra-articular ankle fracture correlate with short- and middle term clinical symptoms after surgery?

Study 3: Does fracture classification and fracture reduction effect clinical outcomes and physical activity?

Method

This study is approved by The National Committee on Health Research Ethics (S-20170139) and The Danish Data Protection Agency (17/28505). Patient recruitment is carried out in the Department of Orthopedic Surgery at Odense University Hospital, Svendborg, while biomarker analyses mainly take places in Department of Neurobiology Research.

All patients diagnosed with intra-articular ankle fracture hospitalized in Odense University Hospital, Svendborg will be recruited to this study.

Prior to surgery synovial fluids are collected from the fracture ankle and contralateral ankle of the same patient. The patient is lying in supine position and the disinfection of both ankles will follow our department's guidelines. A 1.5 x 50 mm needle is inserted in the joint line using the anteromedial or anterolateral approach. Once the needle is in the joint space, a volume of 5.0 ml isotonic saline will be injected in the joint place and mixed before retraction. All patients will have antibiotic coverage prior to surgery to minimize the risk of infection. This procedure is mainly performed by two surgeons (TP and HS), who have great experience in this procedure. In case other surgeons collect the sample, X-ray may be used for assistance. Synovial fluid will be collected, transferred in a 10 ml glass, and within 2 hours transported to the Department of Clinical Biochemistry and Pharmacology for centrifugation and storage at minus 80 degrees celsius. At the end of each month all samples will be transferred in dry ice to the Department of Molecular Endocrinology to be stored in liquid nitrogen. Blood samples will also be collected in Ethylenediaminetetraacetic acid (EDTA) glasses for comparison.

For the discrimination between the fracture and the anterolateral healthy joint, a proteomics analysis is used to identify the classical pro-inflammatory cytokines and the cytokines involving in the extracellular breakdown and cartilage degeneration. For that purpose, a custom multi-ELISA Plex including (IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, tumor necrosis factor (TNF-α), IL-1α, TNF-β, basic fibroblast growth factor (bFGF), IL-1RA), Human matrix metalloproteinase (MMP) 3-Plex Ultra-Sensitive Kit, U-PLEX TGF-β Combo, Aggrecan and CTX-2, will be performed.

The following epidemiological parameters will be recorded: age, sex, body mass index, classification of injury according to Arbeitsgemeinschaft für Osteosynthesefragen (AO) standards, allowed weight bearing, aftercare follows the Odense guidelines with a static walker. All patients will be evaluated at 3 and 12 months post injury according to the following clinical parameters:

Pain (visual analog scale), return to work (days), swelling (measurement of circumference at malleoli (cm)), ankle X-ray, 3D-rotational tomography, 7 days activity tracking and validated scores (the American Orthopedic Foot and Ankle Score (AOFAS), the Foot Function Index - DK (FFI.DK), the Euroqol 5D questionnaire (EQ5D).To reach a power of 80 %, we include 62 patients in our study. Because no previous studies have compared level of pro-inflammatory cytokines with clinical scores, the power estimation is based on a very high standard deviation, loss of follow-up and clinical importance. The investigators plan to perform an interim analysis, when a number of 40 patients is reached.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Existence of an acute fracture involving the ankle (location AO43,AO44) requiring open or closed reduction and internal or external fixation within 14 days
* Being able to read and understand Danish
* Informed consent

Exclusion Criteria:

* Open fractures
* Associated arterial and nerve injuries
* Multiple injured patients with an Injury Severity Score >16
* Primary or secondary infections
* Injuries associated to a Charcot foot
* Signs of existing OA on X-ray

  * Others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients hospitalize in Odense University, Svendborg (31th. Oct. 2017-Jan. 2019) will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of cytokines in fracture ankle versus non-fracture ankle | During surgery
  Multiplex ELISA kits will be use to identify cytokines in both ankles. Cytokines with significant difference will be identified.
Cytokines (identified in primary outcome 1) correlation with clinical outcomes (AOFAS) | 12 months after surgery
  The identified cytokines in the fracture ankle (fracture non fracture ratio above 2.0) will be coupled to the scores of functional foot score (AOFAS), The American Orthopedic Foot and Ankle Score, includes pain, function, alignment, for AOFAS calculation the subscores are added, ranges between 0 (worst) and 100 (best) points

SECONDARY OUTCOMES:
Cytokines (identified in primary outcome 1) correlation with clinical outcomes (FFI.DK) | 12 months after surgery
  The identified cytokines in the fracture ankle (fracture non fracture ratio above 2.0) will be coupled to the scores of FFI.DK, a functional foot score
Cytokines (identified in primary outcome 1) correlation with clinical outcomes (EQ5D-5L) | 12 months after surgery
  The identified cytokines in the fracture ankle (fracture non fracture ratio above 2.0) will be coupled to the scores of EQ5D-5L
Cytokines (identified in primary outcome 1) correlation with clinical outcomes (VAS-score) | 12 months after surgery
  The identified cytokines in the fracture ankle (fracture non fracture ratio above 2.0) will be coupled to VAS-score, a Visual Analog Scale.VAS 0 (best) - 10 (worst)
Cytokines (identified in primary outcome 1) correlation with clinical outcomes (Swelling) | 12 months after surgery
  The identified cytokines in the fracture ankle (fracture non fracture ratio above 2.0) will be coupled to swelling, difference in fracture and non-fracture ankle, measured in millimeters
Cytokines (identified in primary outcome 1) correlation with clinical outcomes (FFI.DK) | 3 months after surgery
  The identified cytokines in the fracture ankle (fracture non fracture ratio above 2.0) will be coupled to the scores of FFI.DK, a functional foot score
Cytokines (identified in primary outcome 1) correlation with clinical outcomes (EQ5D-5L) | 3 months after surgery
  The identified cytokines in the fracture ankle (fracture non fracture ratio above 2.0) will be coupled to the scores of EQ5D-5L
Cytokines (identified in primary outcome 1) correlation with clinical outcomes (VAS-score) | 3 months after surgery
  The identified cytokines in the fracture ankle (fracture non fracture ratio above 2.0) will be coupled to the scores of VAS-score, a Visual Analog Scale.VAS 0 (best) - 10 (worst)
Cytokines (identified in primary outcome 1) correlation with clinical outcomes (Swelling) | 3 months after surgery
  The identified cytokines in the fracture ankle (fracture non fracture ratio above 2.0) will be coupled to swelling, difference in fracture and non-fracture ankle, measured in millimeters

OTHER OUTCOMES:
Correlation between fracture classification and clinical outcomes (AOFAS) | 12 months after surgery
  Fracture classification on pre-operative X-ray (AO classification, 43A, 43B, 43C, 44A, 44B,44C), will be correlated to the scores of functional foot score (AOFAS), The American Orthopedic Foot and Ankle Score, includes pain, function, alignment, for AOFAS calculation the subscores are added, ranges between 0 (worst) and 100 (best) points
Correlation between fracture classification and clinical outcomes (FFI.DK) | 12 months after surgery
  Fracture classification on pre-operative X-ray (AO classification, 43A, 43B, 43C, 44A, 44B,44C), will be correlated to the scores of functional foot score (FFI.DK)
Correlation between fracture classification and clinical outcomes (EQ5D-5L) | 12 months after surgery
  Fracture classification on pre-operative X-ray (AO classification, 43A, 43B, 43C, 44A, 44B,44C), will be correlated to the scores of EQ5D-5L
Correlation between fracture classification and clinical outcomes (VAS-score) | 12 months after surgery
  Fracture classification on pre-operative X-ray (AO classification, 43A, 43B, 43C, 44A, 44B,44C), will be correlated to the scores of VAS-score, a Visual Analog Scale.VAS 0 (best) - 10 (worst)
Correlation between fracture classification and clinical outcomes (Swelling) | 12 months after surgery
  Fracture classification on pre-operative X-ray (AO classification, 43A, 43B, 43C, 44A, 44B,44C), will be correlated to swelling, difference in fracture and non-fracture ankle, measured in millimeters
Correlation between fracture classification and clinical outcomes (activity) | 12 months after surgery
  Fracture classification on pre-operative X-ray (AO classification, 43A, 43B, 43C, 44A, 44B,44C), will be correlated to activity, meassured with an activity tracker, recording number of active minutes per day
Correlation between fracture reduction and clinical outcomes (AOFAS) | 12 months after surgery
  Fracture reduction with conventional X-ray and 3D-rotation CT (e.g. step-off>2 mm, tibiotalartilt >2° and deviation of rotation > 6°) will be correlated to the scores of functional foot score (AOFAS), The American Orthopedic Foot and Ankle Score, includes pain, function, alignment, for AOFAS calculation the subscores are added, ranges between 0 (worst) and 100 (best) points
Correlation between fracture reduction and clinical outcomes (FFI.DK) | 12 months after surgery
  Fracture reduction with conventional X-ray and 3D-rotation CT (e.g. step-off>2 mm, tibiotalartilt >2° and deviation of rotation > 6°) will be correlated to the scores of functional foot score (FFI.DK)
Correlation between fracture reduction and clinical outcomes (EQ5D-5L) | 12 months after surgery
  Fracture reduction with conventional X-ray and 3D-rotation CT (e.g. step-off>2 mm, tibiotalartilt >2° and deviation of rotation > 6°) will be correlated to the scores of EQ5D-5L
Correlation between fracture reduction and clinical outcomes (VAS-score) | 12 months after surgery
  Fracture reduction with conventional X-ray and 3D-rotation CT (e.g. step-off>2 mm, tibiotalartilt >2° and deviation of rotation > 6°) will be correlated to the scores of VAS-score, a Visual Analog Scale.VAS 0 (best) - 10 (worst)
Correlation between fracture reduction and clinical outcomes (Swelling) | 12 months after surgery
  Fracture reduction with conventional X-ray and 3D-rotation CT (e.g. step-off>2 mm, tibiotalartilt >2° and deviation of rotation > 6°) will be correlated to swelling, difference in fracture and non-fracture ankle, measured in millimeters
Correlation between fracture reduction and clinical outcomes (activity) | 12 months after surgery
  Fracture reduction with conventional X-ray and 3D-rotation CT (e.g. step-off>2 mm, tibiotalartilt >2° and deviation of rotation > 6°) will be correlated to activity, meassured with an activity tracker, recording number of active minutes per day

CONTACTS AND LOCATIONS:
Overall Officials: Søren Overgaard, Professor, Principal Investigator — The Orthopaedic Research Unit
Locations (1):
- The Orthopaedic Research Unit, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pham TM, Kristiansen EB, Frich LH, Lambertsen KL, Overgaard S, Schmal H. Association of acute inflammatory cytokines, fracture malreduction, and functional outcome 12 months after intra-articular ankle fracture-a prospective cohort study of 46 patients with ankle fractures. J Orthop Surg Res. 2021 May 25;16(1):338. doi: 10.1186/s13018-021-02473-8. PMID 34034772
- [Derived] Pham TM, Frich LH, Lambertsen KL, Overgaard S, Schmal H. Elevation of Inflammatory Cytokines and Proteins after Intra-Articular Ankle Fracture: A Cross-Sectional Study of 47 Ankle Fracture Patients. Mediators Inflamm. 2021 Jan 8;2021:8897440. doi: 10.1155/2021/8897440. eCollection 2021. PMID 33505222